CLINICAL TRIAL: NCT07026500
Title: A Single-center, Randomized, Double-blind Clinical Trial to Evaluate the Safety and Batch Consistency of the EV71 Vaccine in Infants Aged 6 to 35 Months After Vaccination According to a Two-dose Immunization Schedule
Brief Title: Clinical Trial for Batch Consistency of EV71 Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-EV71-4009; CTR20191800 (Other: China National Medical Products Administration)
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: EV71 Vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Batch group 1 (Experimental): EV71 vaccine first commercial production batch
  Interventions: Biological: EV71 Vaccine
- Batch group 2 (Experimental): EV71 vaccine second commercial production batch
  Interventions: Biological: EV71 Vaccine
- Batch group 3 (Experimental): EV71 vaccine third commercial production batch
  Interventions: Biological: EV71 Vaccine

INTERVENTIONS:
Biological: EV71 Vaccine — EV71 vaccine of commercial production batch

SUMMARY:
This trial is designed as a single-center, randomized, double-blind study. A total of 720 infants aged 6 to 35 months are selected (with 240 subjects in each age group: 6-11 months, 12-23 months, and 24-35 months). Subjects from different age groups are randomly allocated to three batch groups in a 1:1:1 ratio, and receive two doses of the EV71 vaccine from the commercial production batch on days 0 and 30. After each vaccination dose, subjects will be observed for immediate reactions for 30 minutes and for solicited adverse events for the next 7 days, as well as for unsolicited adverse events over the 30 days following vaccination. All subjects will have blood samples collected on day 0 (pre-immunization) and day 60 for serum antibody testing. Additionally, 270 subjects will be selected, for additional blood sampling at various time points: 7 days, 14 days, and 30 days after the first dose, and 7 days and 14 days after the second dose, to assess the EV71 antibody levels at different timepoints following various doses of vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Infants and young children aged 6 to 35 months.
* Able to provide legal identification.
* The guardian of the subject has the ability to understand and agrees to sign the informed consent form.

Exclusion Criteria:

* Previous vaccination with the EV71 vaccine.
* History of hand, foot, and mouth disease.
* History of allergies, asthma, including allergies to vaccines or vaccine components, and severe adverse reactions to vaccines, such as urticaria, difficulty breathing, angioedema, or abdominal pain.
* Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.
* Autoimmune diseases or immune deficiencies/immunosuppression.
* Severe neurological disorders (epilepsy, convulsions, or seizures) or mental illness.
* History of thyroidectomy, asplenia, functional asplenia, or any condition leading to asplenia or splenectomy.
* Blood coagulation abnormalities diagnosed by a physician (such as clotting factor deficiencies, coagulopathies, platelet abnormalities) or evident bruising or bleeding disorders.
* Treatment with immunosuppressants, cytotoxic therapy, or inhaled corticosteroids within 6 months prior to enrollment (excluding corticosteroid nasal spray therapy for allergic rhinitis, or topical corticosteroid treatment for acute non-complicated dermatitis).
* Receipt of blood products within 3 months prior to vaccination with the trial vaccine.
* Receipt of other investigational vaccines within 30 days prior to vaccination with the trial vaccine.
* Receipt of live attenuated vaccines within 14 days prior to vaccination with the trial vaccine.
* Receipt of subunit or inactivated vaccines within 7 days prior to vaccination with the trial vaccine.
* Any acute illness or acute exacerbation of chronic illness within the past 7 days.
* Fever before receiving the investigational vaccine, with an axillary temperature > 37.0°C.
* Any other factors that, in the investigator's judgment, make the subject unsuitable for participation in the clinical trial.

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 720 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
The GMT of EV71 neutralizing antibodies 30 days after complete immunization with the EV71 vaccine | 30 days after second dose

SECONDARY OUTCOMES:
Seroconversion rates, seropositive rates, and GMT of antibodies at 7 days, 14 days, and 30 days after the first dose of the EV71 vaccine | 7,14 and 30 days after the first dose
Seroconversion rates, seropositive rates, and GMT of antibodies at 7 days and 14 days after the second dose of the EV71 vaccine, as well as the seroconversion rate and seropositive rate at 30 days post-vaccination | 7,14 and 30 days after the second dose
The incidence of adverse reactions within 30 days after each dose of the EV71 vaccine | 30 days after each dose
The incidence of solicited adverse events within 0-7 days after each dose of the EV71 vaccine | 7 days after each dose
The incidence of serious adverse events during the safety observation period | 30 days after the second dose

CONTACTS AND LOCATIONS:
Locations (1):
- Dazhu County Center for Disease Control and Prevention, Dazhu, China

IPD SHARING:
Plan to Share IPD: No